CLINICAL TRIAL: NCT05542368
Title: Study of Thyroid State in Patients With Inflammatory Bowel Diseases
Brief Title: Study of Thyroid Status in Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesreen Hassan Mansour Ali, Principal Investigator, Assiut University
Other Study IDs: thyroid state in IBD patients
Record Dates: First submitted 2022-05-20; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Thyroid Disease; Irritable Bowel Disease
MeSH Terms: conditions — Thyroid Diseases; Irritable Bowel Syndrome | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with IBD: All patients were subjected to history taking and physical examination with emphasis on history of autoimmune disease, extraintestinal manifestations of IBD, neck examination for goiter, symptoms and signs of thyroid dysfunction.
  b) Laboratory investigations: Thyroid function test (include T3-T4- TSH)
  * ESR - CRP - thyroid antibodies: (Anti TPO -Anti Thyroglobulin)
    c)-Imaging:
  * Neck U/S on thyroid gland to identify patients with ultrasonographic evidence of autoimmune thyroiditis (diffuse hypoechogenicity or heterogenicity echotexture or both) and to detect thyroid nodularity.
  d ) Endoscopic findings regarding diagnosis of IBD confirmed by histopathological examination
  Interventions: Diagnostic Test: Thyroid tests
- Healty individuals as a control group: All patients were subjected to history taking and physical examination with emphasis on history of autoimmune disease, extraintestinal manifestations of IBD, neck examination for goiter, symptoms and signs of thyroid dysfunction.
  b) Laboratory investigations: Thyroid function test (include T3-T4- TSH)
  * ESR - CRP - thyroid antibodies: (Anti TPO -Anti Thyroglobulin)
    c)-Imaging:
  * Neck U/S on thyroid gland to identify patients with ultrasonographic evidence of autoimmune thyroiditis (diffuse hypoechogenicity or heterogenicity echotexture or both) and to detect thyroid nodularity.
  Interventions: Diagnostic Test: Thyroid tests

INTERVENTIONS:
Diagnostic Test: Thyroid tests — Thyroid function test TSH ,T3,T4 Thyroid antibody test anti TPO,antithyroglobulin
  Other Names: Thyroid function test and thyroid antibodies

SUMMARY:
. The aim of the present study is to study thyroid state in patients with IBD

DETAILED DESCRIPTION:
All patients were subjected to history taking and physical examination with emphasis on history of autoimmune disease, extraintestinal manifestations of IBD, neck examination for goiter, symptoms and signs of thyroid dysfunction.

b) Laboratory investigations: Thyroid function test (include T3-T4- TSH)

* ESR - CRP - thyroid antibodies: (Anti TPO -Anti Thyroglobulin)

  c)-Imaging:
* Neck U/S on thyroid gland to identify patients with ultrasonographic evidence of autoimmune thyroiditis (diffuse hypoechogenicity or heterogenicity echotexture or both) and to detect thyroid nodularity.

d ) Endoscopic findings regarding diagnosis of IBD confirmed by histopathological examination

ELIGIBILITY:
Inclusion Criteria: All patients with IBD

-

Exclusion Criteria:

* patients with
* Thyroid disease
* Acute or chronic kidney
* Acute or Chronic Liver Disease. Active Lupus -
* Malignancy
* patients taking medications that affect thyroid function as rifampin, amiodarone …..

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with IBD admitted at Assiut University Hospital, Al Rajhi Liver Hospital or attending IBD outpatient clinic.
  a. Inclusion criteria: All patients with IBD Exclusion criteria: patients with
  * Thyroid disease
  * Acute or chronic kidney
  * Acute or Chronic Liver Disease. Active Lupus -
  * Malignancy
  * patients taking medications that affect thyroid function as rifampin, amiodarone
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of thyroid disorders in patients with IBD | 1 year
  By use of Thyroid function test (include T3-T4- TSH), thyroid antibodies and thyroid sonography

CONTACTS AND LOCATIONS:
Overall Officials: Abo zaid Ali, assistant prof, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: nflammatory bowel disease severity and activity are correlated to thyroid gland nodularity, chronic nonthyroidal illness, and thyroid autoantibodies but not thyroid dysfunction — https://www.ejode.eg.net/article.asp?issn=2356-8062;year=2016;volume=2;issue=2;spage=67;epage=80;aulast=Ghitany
- See also: Role of autoantibodies in the pathogenesis and association of endocrine autoimmune disorders — http://pubmed.ncbi.nlm.nih.gov/3065074
- See also: Autoimmune thyroid disease (Graves' disease and hashimoto's thyroiditis) in two patients with Crohn's disease: case reports and literature review — https://pubmed.ncbi.nlm.nih.gov/15897640/
- See also: Simultaneous occurrence of inflammatory bowel disease and thyroid disease — https://pubmed.ncbi.nlm.nih.gov/11419852/
- See also: Coexistence of Addison's disease, ulcerative colitis, hypothyroidism and pernicious anemia — https://pubmed.ncbi.nlm.nih.gov/1500669/